CLINICAL TRIAL: NCT00000546
Title: Stress Reduction and Atherosclerotic CVD in Blacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 90; R01HL051519 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases; Coronary Disease | interventions — Meditation

INTERVENTIONS:
Behavioral: meditation

SUMMARY:
To evaluate the effectiveness of stress reduction with Transcendental Meditation (TM) on left ventricular hypertrophy, left ventricular function, blood pressure, psychosocial stress and quality of life, and cardiovascular disease risk factors.

DETAILED DESCRIPTION:
BACKGROUND:

Blacks in the United States have disproportionately high rates of cardiovascular disease and mortality. Left ventricular hypertrophy, the primary manifestation of hypertensive heart disease and a major independent predictor of cardiovascular mortality, is twice as prevalent in Blacks with hypertension as in whites. Research has implicated chronic socio-environmental and psychological stress in the etiology of hypertension and left ventricular hypertrophy in Blacks. The trial seeks to investigate directly the impact of stress reduction programs for treating hypertensive heart disease in Blacks, since conventional antihypertensive drug therapies are less successful than expected. Moreover, these therapies frequently have adverse side effects on quality of life, and have low compliance rates, particularly in minorities.

DESIGN NARRATIVE:

The first study conducted between 1994 and 1999 used transcendental meditation for stress reduction in hypertensive heart disease. The study was randomized and blind. Subjects were randomized to practice TM for twelve months or to receive health education. The following measurements were obtained: left ventricular mass and function using echocardiography; clinic blood pressure and ambulatory blood pressure monitoring; urinary sodium excretion; alcohol consumption, weight, physical activity, cigarette smoking, and previous use of antihypertensive medication; various quality of life measures including physical functioning, psychosocial functioning, subjective symptoms, trait anger and anger-expression, stress impact scale, personal efficacy and health locus of control, social supports, ego development, and social desirability.

The trial was part of the Collaborative Projects on Minority Health, an Institute- initiated program to foster collaborative clinical research that focused on new and improved approaches for diagnosis, management, and prevention of cardiovascular, lung, and blood diseases in minorities. The trial was part of a two-grant collaboration on Nonpharmacologic Treatments for Managing Hypertension in African American Adults. Ernest Johnson (R01HL50516),the Program Coordinator collaborated with Robert Schneider (R01HL51519). The objectives of their studies were complementary and the collaborative arrangements allowed them to determine the effectiveness of different approaches to stress management in comparison with a control group that was comparable at both sites. In addition, the treatment schedules in both studies resulted in identical contact time, length of interventions, expectations regarding treatment effectiveness, and follow-up assessment periods. As a result, a considerable degree of pooling of data for analysis was possible.

Dr. Schneider's study was renewed in FY 1999 to conduct a randomized, single-blind, controlled, community-based trial involving 184 African American subjects with known coronary heart disease. Male and female subjects are enrolled at the on-going field site, Martin Luther King-Drew Medical Center in inner city Los Angeles. After baseline testing, subjects are randomized to either active stress reduction with TM or health education control-both in addition to usual medical care-and posttested after 12 months. The primary outcome is carotid artery atherosclerosis (IMT) measured non-invasively by quantitative B-mode ultrasonography. Secondary measures include traditional CVD risk factors (blood pressure, lipids, smoking, exercise), psychosocial stress, quality of life and cost effectiveness.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-03; Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schneider — Maharishi International University

REFERENCES:
- [Background] Schneider RH, Castillo-Richmond A, Alexander CN, Myers H, Kaushik V, Aranguri C, Norris K, Haney C, Rainforth M, Calderon R, Nidich S. Behavioral treatment of hypertensive heart disease in African Americans: rationale and design of a randomized controlled trial. Behav Med. 2001 Summer;27(2):83-95. doi: 10.1080/08964280109595775. PMID 11763829
- [Background] Castillo-Richmond A, Schneider RH, Alexander CN, Cook R, Myers H, Nidich S, Haney C, Rainforth M, Salerno J. Effects of stress reduction on carotid atherosclerosis in hypertensive African Americans. Stroke. 2000 Mar;31(3):568-73. doi: 10.1161/01.str.31.3.568. PMID 10700487
- [Background] Calderon R Jr, Schneider RH, Alexander CN, Myers HF, Nidich SI, Haney C. Stress, stress reduction and hypercholesterolemia in African Americans: a review. Ethn Dis. 1999 Autumn;9(3):451-62. PMID 10600068